CLINICAL TRIAL: NCT02855086
Title: Open-Label Study Evaluating Cetuximab-IRDye800 as an Optical Imaging Agent to Detect Neoplasms During Neurosurgical Procedures
Brief Title: Cetuximab-IRDye 800CW in Detecting Tumors in Patients With Malignant Glioma Undergoing Surgery
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: logistics
Sponsor: Eben Rosenthal (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Eben Rosenthal, Professor of Otolaryngology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-37595; NCI-2016-01165 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRNCNS0008 (Other: Stanford Cancer Institute); P30CA124435 (NIH); IRB-37595 (Other: Stanford IRB)
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Brain Neoplasm; Malignant Glioma
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Cetuximab; Antibodies, Monoclonal; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 50 mg cetuximab-IRDye 800 (Experimental): Patients receive cetuximab IV over 30 minutes and a lower dose of cetuximab IRDye800 IV over 30 minutes to 1 hour on day 0.
  All patients undergo standard of care surgical resection of tumor on days 2 to 5.
  Interventions: Biological: Cetuximab; Drug: Cetuximab-IRDye 800CW; Procedure: Tumor resection
- 100 mg cetuximab-IRDye 800 (Experimental): Patients receive cetuximab IV over 30 minutes and a higher dose of cetuximab IRDye800 IV over 30 minutes to 1 hour on day 0.
  All patients undergo standard of care surgical resection of tumor on days 2 to 5.
  Interventions: Biological: Cetuximab; Drug: Cetuximab-IRDye 800CW; Procedure: Tumor resection

INTERVENTIONS:
Biological: Cetuximab — Administered intravenously (IV)
  Other Names: Erbitux; Chimeric Anti-epidermal growth factor receptor (EGFR0 monoclonal antibody; Chimeric Monoclonal Antibody (MoAb) C225; IMC-C225
Drug: Cetuximab-IRDye 800CW — Administered intravenously (IV)
  Other Names: Cetuximab-IRDye 800; Cetuximab-IRDye800; Cetuximab-IRDye800CW
Procedure: Tumor resection — Standard of care treatment
  Other Names: Conventional Surgery

SUMMARY:
This study is a phase 1-2 trial that evaluates the best dose of cetuximab-IRDye 800CW and how well it works in detecting tumors in patients with malignant glioma who are undergoing surgery. Cetuximab-IRDye 800CW is an optical imaging agent that may help detect tumor cells when a special camera is used.

DETAILED DESCRIPTION:
This is a dose-escalation study of cetuximab-IRDye 800CW. Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive cetuximab intravenously (IV) over 30 minutes and a lower dose of cetuximab IRDye800 IV over 30 minutes to 1 hour on day 0.

COHORT II: Patients receive cetuximab IV over 30 minutes and a higher dose of cetuximab IRDye800 IV over 30 minutes to 1 hour on day 0.

All patients undergo standard of care surgical resection of tumor on days 2-5.

After completion of study, patients are followed up at days 10 and 30.

PRIMARY OBJECTIVE:

Determine the efficacy of cetuximab-IRDye 800CW (cetuximab IRDye800) in intraoperatively identifying malignant glioma compared to surrounding normal central nervous system tissue, as measured by tumor-to-background ratio.

SECONDARY OBJECTIVE:

Determine the tolerability of the cetuximab IRDye800 as an imaging agent in subjects undergoing resection of malignant glioma.

ELIGIBILITY:
INCLUSION CRITERIA

* Suspected brain tumors to undergo removal (surgical resection) as standard of care, as assessed by the operating surgeon
* Life expectancy of > 12 weeks
* Karnofsky performance status of at least 70% or Eastern Cooperative Oncology Group (ECOG)/Zubrod level 1
* Hemoglobin ≥ 9 gm/dL
* Platelet count ≥ 100,000/mm³
* Magnesium, potassium and calcium > the lower limit of normal per institution normal lab values
* Thyroid-stimulating hormone (TSH) < 13 micro international units/mL

EXCLUSION CRITERIA

* Received an investigational drug within 30 days prior to first dose of cetuximab IRDye800
* Within 6 months prior to enrollment, myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina
* History of infusion reactions to cetuximab or other monoclonal antibody therapies
* Evidence of QT prolongation on pretreatment electrocardiogram (ECG) (greater than 440 ms in males or greater than 450 ms in females)
* Receiving class IA (quinidine, procainamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-11-08 (Actual); Study Completion 2016-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Li, MD, Principal Investigator — Stanford University; Eben Rosenthal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Cetuximab, Lower Dose Cetuximab-IRDye 800, Surgery): Patients receive cetuximab IV over 30 minutes and a lower dose of cetuximab IRDye800 IV over 30 minutes to 1 hour on day 0.
  All patients undergo standard of care surgical resection of tumor on days 2 to 5.
  Cetuximab: Given IV
  Cetuximab-IRDye 800CW: Given IV
  Conventional Surgery: Undergo tumor resection
  Laboratory Biomarker Analysis: Correlative studies
- Cohort 2 (Cetuximab, Higher Dose Cetuximab-IRDye 800, Surgery): Patients receive cetuximab IV over 30 minutes and a higher dose of cetuximab IRDye800 IV over 30 minutes to 1 hour on day 0.
  All patients undergo standard of care surgical resection of tumor on days 2 to 5.
  Cetuximab: Given IV
  Cetuximab-IRDye 800CW: Given IV
  Conventional Surgery: Undergo tumor resection
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Cohort 1 (Cetuximab, Lower Dose Cetuximab-IRDye 800, Surgery) | Cohort 2 (Cetuximab, Higher Dose Cetuximab-IRDye 800, Surgery)
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Cetuximab, Lower Dose Cetuximab-IRDye 800, Surgery) | Cohort 2 (Cetuximab, Higher Dose Cetuximab-IRDye 800, Surgery) | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Tumor to Background Ratio (TBR)
Description: Tumor to background ratios (TBR) will be generated from still images by comparing the relative fluorescence of normal and tumor tissue. The average fluorescence will be compared to the average fluorescence of the surrounding tissue using the paired student's T test for each specimen.
Time Frame: 1 day
Measure: Mean (Full Range); unit: Fluorescence Tumor to background ratio
Arm/Group | Cohort 1 (Cetuximab, Lower Dose Cetuximab-IRDye 800, Surgery) | Cohort 2 (Cetuximab, Higher Dose Cetuximab-IRDye 800, Surgery)
Number analyzed (Participants) | 2 | 1
Fluorescence Tumor to background ratio | 1.39 [1.20 to 1.58] | 2.65 [2.65 to 2.65]

2. Secondary Outcome: Incidence of Adverse Events
Description: The incidence of serious and non-serious adverse events is reported as the number of adverse events (Grade 2 or higher), as graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Data are reported by number of events by treatment level.
Time Frame: Up to 30 days
Measure: Number; unit: Adverse events
Arm/Group | Cohort 1 (Cetuximab, Lower Dose Cetuximab-IRDye 800, Surgery) | Cohort 2 (Cetuximab, Higher Dose Cetuximab-IRDye 800, Surgery)
Number analyzed (Participants) | 2 | 1
Adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Cohort 1 (Cetuximab, Lower Dose Cetuximab-IRDye 800, Surgery) | Cohort 2 (Cetuximab, Higher Dose Cetuximab-IRDye 800, Surgery)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Cetuximab, Lower Dose Cetuximab-IRDye 800, Surgery) (N=2) | Cohort 2 (Cetuximab, Higher Dose Cetuximab-IRDye 800, Surgery) (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Nervous system disorders - Other, Imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No